CLINICAL TRIAL: NCT06697626
Title: Food4PD: Validation of a Novel Functional Food Designed to Meet the Nutritional Needs of People Living With Parkinson's
Brief Title: Validation of a Novel Functional Food Designed to Meet the Nutritional Needs of People Living With Parkinson's Disease
Acronym: Food4PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: University of Leeds (Other); University of Auckland, New Zealand (Other); Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC/24/0034
Record Dates: First submitted 2024-11-15; First posted 2024-11-20 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2024-11

CONDITIONS: Constipation; Parkinson Disease
Keywords: Constipation; Fibre; B-vitamins; Functional food; Nutritional status; Parkinson disease
MeSH Terms: conditions — Constipation; Parkinson Disease | interventions — Inulin; Folic Acid; Vitamin D

STUDY DESIGN:
Intervention Model Description: Twice daily intervention for 12 weeks with one of the following treatments (in powder form):
  1. An enriched functional drink containing chicory inulin (10g), folic acid (100µg), vitamin B12 (5µg), vitamin B6 (5mg), riboflavin (2.5mg) and vitamin D (5µg).
  2. A control/placebo drink with similar energy content but without the additional nutrient provision.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dietary Supplement (Functional drink) (Active Comparator): An enriched functional drink containing chicory inulin (10g), folic acid (100µg), vitamin B12 (5µg), vitamin B6 (5mg), riboflavin (2.5mg) and vitamin D (5µg).
  This drink will be consumed twice daily for an intervention period of 12 weeks
  Interventions: Dietary Supplement: Inulin, B-vitamins and vitamin D
- Placebo drink (Placebo Comparator): A placebo drink drink with similar energy content but without the additional nutrient provision.
  This drink will be consumed twice daily an intervention period of 12 weeks.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Inulin, B-vitamins and vitamin D — Intervention twice daily with:
  10g chicory inulin 100µg folic acid 5µg vitamin B12 5mg vitamin B6 2.5mg riboflavin 5µg vitamin D
  Arms: Dietary Supplement (Functional drink)
Dietary Supplement: Placebo group — A twice daily placebo drink with similar energy content but without the additional nutrient provision
  Arms: Placebo drink

SUMMARY:
Constipation is a common complication and non-motor symptom of Parkinson's disease (PD) and affects up to 80% of people with PD. It is in fact within the non-motor symptoms that nutrition and dietetic intervention could have the greatest impact. Research suggests that increasing the amount of fibre in the diet could help to alleviate the effects of constipation. Inulin is a type of fibre widely found in a variety of vegetables, and recent studies have shown that inulin can improve constipation in people with PD. With the assistance of a food company, the investigators have developed a functional drink, enriched with chicory inulin and other key nutrients, including B-vitamins and vitamin D (which are suggested within the literature to be beneficial in PD). Therefore, the investigators plan to conduct a 12-week feasibility study to test the effect of this novel functional drink on gut health outcomes, nutritional status, and overall quality of life in people living with PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson Disease (PD)
* Aged ≥18 years
* Individuals with the capacity to provide informed consent

Exclusion Criteria:

* Individuals with PD living in institutional care or in hospital
* Drug, infection or toxin induced parkinsonism
* Individuals with diabetes
* B12 injection users
* Currently taking antibiotics
* Using supplements containing the nutrients of interest (B-vitamins, inulin, probiotics)
* Any other medical, cognitive or psychosocial issue, or co-enrolment in another study, that could interfere or disrupt adherence to the study requirements
* An allergy to any of the ingredients in the functional and/or control drinks
* Consuming a fermented food and/or probiotic yogurts on a daily basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All
Enrollment: 56 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Dietary fibre intake | 12 weeks
  A food frequency questionnaire and 4-day food diary will be completed and analysed using nutritional analysis software to determine intake of dietary fibre (g/day) pre- and post- intervention.
Gut microbiome profile | 12 weeks
  Faecal samples will be collected to examine the gut microbiome profile using faecal 16S rRNA profiling, V3-V4 region and QIIME2 pipeline.
Quality of life assessment | 12 weeks
  Assessed using The Parkinson's Disease Questionnaire (PDQ-39). This 39-item questionnaire assesses how often participants with Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication. Answers are based on a 5-point ordinal scoring system ranging from 0 to 4, with lower scores reflecting a better quality of life.
Parkinsons Disease symptoms | 12 weeks
  Assessed using the MDS-Unified Parkinson Disease Rating Scale (MDS-UDPRS). The MDS-UPDRS has four parts: I: Non-motor Experiences of Daily Living; II: Motor Experiences of Daily Living; III: Motor Examination; IV: Motor Complications. Each question is anchored with five responses that are linked to commonly accepted clinical terms: 0=normal, 1=slight, 2=mild, 3=moderate, and 4=severe. Higher scores indicate more severe impairment.
Gastrointestinal symptoms | 12 weeks
  Assessed using the Gastrointestinal Symptom Rating Scale. This 15-item questionnaire uses a seven-graded Likert scale, where 1 represents the most positive option and 7 the most negative option. Higher scores indicate more severe symptoms.
Constipation | 12 weeks
  Assessed using the Bristol Stool Chart, a diagnostic tool that participants can use to classify their stools based on their appearance. The chart ranges from type 1 (hard) to type 7 (loose, watery) and may identify problems with bowel movements through the shape and consistency of the stool.

SECONDARY OUTCOMES:
Vitamin B12 | 12 weeks
  Serum total vitamin B12 measured by microbiological assay based on a colistin sulphate-resistant strain of Lactobacillus leichmannii; serum methylmalonic acid measured by gas chromatography-tandem mass spectrometry based on methylchloroformate derivatisation.
Folate | 12 weeks
  Serum folate and red blood cell folate measured by microbiological assay based on a chloramphenicol-resistant strain of Lactobacillus casei.
Vitamin B6 | 12 weeks
  Vitamin B6 status as measured by plasma pyridoxal-5-phosphate using high-performance liquid chromatography with fluorescence detection.
Riboflavin | 12 weeks
  Measured using the functional assay erythrocyte glutathione reductase activation coefficient, EGRac
Serum total homocysteine | 12 weeks
  Measured by gas chromatography-tandem mass spectrometry based on methylchloroformate derivatisation.
Vitamin D | 12 weeks
  Vitamin D as measured by serum 25-hydroxyvitamin D status, using liquid chromatography mass spectrometry.
Inflammation | 12 weeks
  Markers of inflammation (analysed by enzyme-linked immunosorbent assay): C-reactive protein (CRP), interleukin 6 (IL-6), interleukin 10 (IL-10), tumour necrosis factor (TNF-α).

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, County Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No